CLINICAL TRIAL: NCT03818308
Title: Multicenter Trial for the Treatment of Acute Hepatitis C for 8 Weeks With Sofosbuvir/Velpatasvir Fix Dose combination_The HepNet Acute HCV-V Study
Brief Title: Trial for the Treatment of Acute Hepatitis C for 8 Weeks With Sofosbuvir/Velpatasvir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: HepNet Study House, German Liverfoundation (Network); Gilead Sciences (Industry); German Center for Infection Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HepNet-aHCV-V; 2018-003474-27 (EudraCT Number)
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C; Acute Hepatitis C
Keywords: Acute hepatitis C virus (HCV) infection
MeSH Terms: conditions — Hepatitis C; Infections | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, single-arm multicenter, phase II pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sofosbuvir and Velpatasvir (Experimental): SOF/VEL FDC film-coated tablet, oral, SOF 400 mg/VEL 100 mg daily, 8 weeks
  Interventions: Drug: Sofosbuvir and Velpatasvir

INTERVENTIONS:
Drug: Sofosbuvir and Velpatasvir — All subjects will receive one film-coated tablet of sofosbuvir/velpatasvir (400/100 mg) orally once daily for 8 weeks.
  Other Names: Epclusa 400 mg/100 mg film-coated tablets

SUMMARY:
This is a single arm multicenter pilot study to evaluate the efficacy and safety of treatment with sofosbuvir (SOF)/velpatasvir (VEL) fix dose combination (FDC) in patients with acute hepatitis C virus (HCV) infection.

DETAILED DESCRIPTION:
This is a single arm multicenter pilot study to evaluate the efficacy and safety of treatment with SOF/VEL FDC for 8 weeks in patients with acute HCV infection as measured by the proportion of subjects with sustained viral response (undetectable HCV RNA) 12 weeks after stop of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Male or female, age > 18 years
3. HCV RNA > 10^3 IU/mL at screening
4. Confirmation of acute HCV infection documented by either:

   1. Documented seroconversion to HCV antibody (anti-HCV) positivity within the 4 months preceding screening
   2. Documented conversion to HCV RNA positivity within the 4 months preceding screening
   3. or known or suspected exposure to HCV within the 4 months preceding screening with 10 times elevated serum ALT level at screening or 4 month preceding screening without evidence of confounding liver disorders
5. Body mass index (BMI) ≥18 kg/m2
6. Subjects must have the following laboratory parameters at screening:

   1. INR ≤ 1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR
   2. HbA1c ≤ 10%
   3. Creatinine clearance (CLcr) ≥ 30 mL/min, as calculated by the Cockcroft-Gault equation (using actual body weight)
7. A negative serum pregnancy test is required for female subjects (unless surgically sterile or women ≥ 54 years of age with cessation for 24 ≥ months of previously occurring menses). Complete abstinence from intercourse. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) is not permitted.

   Or

   Consistent and correct use of 1 of the following methods of birth control listed below, in addition to a male partner who correctly uses a condom, from the date of Screening until the end of follow up:
   * intrauterine device (IUD) with a failure rate of < 1% per year
   * female barrier method: cervical cap or diaphragm with spermicidal agent
   * tubal sterilization
   * vasectomy in male partner
   * hormone-containing contraceptive:

     * implants of levonorgestrel
     * injectable progesterone
     * oral contraceptives (either combined or progesterone only)
     * contraceptive vaginal ring
     * transdermal contraceptive patch
8. Subject must be able to comply with the dosing instructions for study drug administration and be able to complete the study schedule of assessments

Exclusion Criteria:

1. Subject has been treated with any investigational drug or device within 42 days of the Screening visit
2. Co-Infection with HIV
3. Clinically-significant illness (other than HCV) or any other major medical disorder that, in the opinion of the investigator, may interfere with subject treatment, assessment or compliance with the protocol.
4. Solid organ transplantation
5. Gastrointestinal disorder or post-operative condition that could interfere with the absorption of the study drug (for example, gastric bypass or severe ulcerative colitis).
6. Clinical signs of hepatic decompensation (i.e., clinical ascites, encephalopathy or variceal hemorrhage).
7. Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy.
8. Psychiatric hospitalization, suicide attempt, and/or a period of disability as a result of their psychiatric illness within the last 2 years. Subjects with psychiatric illness that is well-controlled on a stable treatment regimen for at least 12 months prior to screening or has not required medication in the last 12 months may be included.
9. Significant drug allergy (such as anaphylaxis or hepatotoxicity).
10. Pregnant or nursing female
11. Clinically-relevant drug or alcohol abuse that significantly impairs patient compliance. Uncontrolled users of intravenous drugs will not be permitted to enroll in the study.
12. Clinical relevant (not controlled) liver disease of a non-HCV etiology (e.g., hemochromatosis, autoimmune hepatitis, alcoholic liver disease, Wilson's disease, α1 antitrypsin deficiency, cholangitis)
13. Use of any prohibited concomitant medications within 21 days before the Baseline/Day 1 visit. The use of amiodarone is prohibited from 60 days prior to Day 1 through the end of treatment;
14. Known hypersensitivity to SOF/VEL or formulation excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with sustained virological response (undetectable HCV RNA) 12 weeks after discontinuation of therapy | 12 weeks after discontinuation of therapy
  Measured by the portion of subjects with sustained virological response (undetectable HCV RNA)

SECONDARY OUTCOMES:
Mean HCV RNA viral load at baseline, 2 weeks, 4 weeks, 8 weeks, and 12 weeks after stop of therapy | at baseline, after 2 weeks, 4 weeks and 8 weeks of therapy, and 12 weeks after stop of therapy
  Measured by mean HCV RNA viral load
Proportion of subjects who reached ALT normalization (ALT < ULN) after 8 weeks of therapy and 12 weeks after discontinuation of therapy | after 8 weeks of therapy, and 12 weeks after discontinuation of therapy
  Measured by the proportion of subjects who reached ALT normalization (ALT < ULN)
Assessment of frequency and severity of adverse events (AEs) | through study completion, an average of 20 weeks
  Collection of all AEs

CONTACTS AND LOCATIONS:
Overall Officials: Markus Cornberg, Prof. Dr., Principal Investigator — Hannover Medical School, Clinic for Gastroenterology, Hepatology, and Endocrinology
Locations (14):
- Germany (14):
  - Zentrum für Infektiologie Prenzlauer Berg, Berlin
  - Charité Campus Virchow-Klinikum, Medizinische Klinik mit Schwerpunkt Hepatologie und Gastroenterologie, Berlin
  - Universitätsklinikum Bonn, Medizinische Klinik und Poliklinik I, Bonn
  - Praxis Hohenstaufenring, Cologne
  - Universitätsklinikum Essen, Klinik für Gastroenterologie und Hepatologie, Essen
  - Klinikum der J.W. Goethe-Universität Frankfurt, Frankfurt
  - Allgemeinmedizinische und internistische Praxis, Friedrichshain
  - Infektionsmedizinisches Centrum Hamburg (ICH) Study Center, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, I. Medizinische Klinik und Poliklinik, Hamburg
  - Medizinische Hochschule Hannover, Innere Medizin, Klinik für Gastroenterologie, Hepatologie und Endokrinologie, Hanover
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Gastroenterologie, Leipzig
  - Klinikum rechts der Isar der TU-München, II Medizinische Klinik und Poliklinik, München
  - Gemeinschaftspraxis - Infectomed, Stuttgart
  - Universitätsklinikum Würzburg, Medizinische Klinik II, Schwerpunkt Infektiologie, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maasoumy B, Ingiliz P, Spinner CD, Cordes C, Stellbrink HJ, Schulze Zur Wiesch J, Schneeweiss SM, Deterding K, Muller T, Kahlhofer J, Dorge P, von Karpowitz M, Manns MP, Wedemeyer H, Cornberg M; HepNet Acute HCV-V Study Group. Sofosbuvir plus velpatasvir for 8 weeks in patients with acute hepatitis C: The HepNet acute HCV-V study. JHEP Rep. 2022 Dec 16;5(3):100650. doi: 10.1016/j.jhepr.2022.100650. eCollection 2023 Mar. PMID 36852107